CLINICAL TRIAL: NCT04379778
Title: Effects of Aerobic Exercise on Brain Health in Parkinson's Disease
Brief Title: Aerobic Exercise and Brain Health in Parkinson's
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Brain Health in Parkinson's
Record Dates: First submitted 2020-04-29; First posted 2020-05-07 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2022-11

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aerobic exercise (Experimental): Moderate to high intensity aerobic exercise for 24 weeks.
  Interventions: Other: Aerobic exercise
- Standard care (No Intervention): Habitual lifestyle including standard care.

INTERVENTIONS:
Other: Aerobic exercise — Progressive moderate to high intensity aerobic exercise.
  Arms: Aerobic exercise

SUMMARY:
The purpose of the project is to investigate how moderate to high intensity aerobic exercise affects brain health in patients with Parkinson's disease. Assessments include MRI, blood markers, cognition, functional tests, questionnaires, and cardiorespiratory fitness.

The study will be a single blinded randomized controlled trial with a 6-month long intervention.

DETAILED DESCRIPTION:
Background: No approved medical treatments preventing, delaying or stopping Parkinson's disease (PD) exist, making identification of interventions having this potential a major priority. Exercise studies have demonstrated beneficial effects of aerobic exercise (AE) on aerobic capacity, cognition, depression and the Unified Parkinson's Disease Rating Scale (UPDRS). Animal studies show that AE can reduce α-synuclein aggregation and toxin-induced lesions in the nigrostriatal pathway while improving motor and cognitive function. Consequently, AE possesses neuroprotective potentials and thus represents a potentially inexpensive and easily accessible disease modifying therapy in PD. Evolving magnetic resonance imaging (MRI) techniques offer valid and reliable biomarkers to monitor disease progression, but no longitudinal MRI study has assessed the neuroprotective potentials of AE in PD.

Aim: To investigate whether 24 weeks of AE can delay PD progression markers and improve motor/non-motor symptoms in PD.

Methods: 70 PD patients will be randomized 1:1 to 24 weeks of supervised AE (60 sessions, moderate to high intensity) or standard care. Neuroprotective effects will be determined by MRI scans (R2*, quantitative susceptibility mapping, diffusion kurtosis imaging, neuromelanin-weighted MRI, volumetry), blood markers and Levodopa equivalents. Clinical (MDS-UPDRS III) and subjective (MDS-UPDRS I) outcomes are also assessed.

Perspectives: By combining expertise from exercise physiology, radiology, endocrinology and neuropsychology a novel approach is taken aiming to understand the possible neuroprotective effects of AE in PD. This would be of high relevance to PD patients and their relatives. From a societal perspective it may lower disability-related costs by optimizing PD rehabilitation. In case of positive findings, this would provide the first convincing human evidence of a disease modifying effect of AE in PD potentially changing clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent
* Age ≥ 40 years
* Idiopathic PD diagnosis (within the previous five years)
* Patients in symptomatic therapy / not in therapy. Patients who are not already taking medication are not expected to need medication within 6 months of inclusion (in case of drug startup, this is noted)
* Hoehn & Yahr ≤ 3
* Ability to transport oneself to and from exercise and testing

Exclusion Criteria:

* Alcohol abuse, depression, pacemaker
* Comorbidity/competing (neurological) disorder preventing participation in the intervention
* Pregnancy
* Metallic implants that prevent MRI.
* Expected exercise adherence below 85% of all planned sessions.
* Systematic moderate-high-level AE more than twice per week prior to start-up in the project

Ages: 40 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2023-10-01 (Actual)

PRIMARY OUTCOMES:
R2* MRI change | 0, 24 and 48 weeks
  Effective transverse relaxation rate (R2*)

SECONDARY OUTCOMES:
QSM MRI change | 0, 24 and 48 weeks
DKI MRI change | 0, 24 and 48 weeks
Neuromelanin MRI change | 0, 24 and 48 weeks
Volumetry MRI change | 0, 24 and 48 weeks
Change in blood markers (e.g. α-synuclein) | 0, 24 and 48 weeks
Change in Levodopa equivalents | 0, 24 and 48 weeks
MDS-UPDRS change | 0, 24 and 48 weeks
Aerobic capacity (VO2max test) | 0, 24 and 48 weeks
Timed up and go (TUG) change | 0, 24 and 48 weeks
6 min walk test (6MWT) change | 0, 24 and 48 weeks
Balance (Mini BESTest) change | 0, 24 and 48 weeks
Cognition (The Montreal Cognitive Assessment (MoCA)) change | 0, 24 and 48 weeks
Health-related quality of life (Parkinson's Disease Questionnaire (PDQ-39)) change | 0, 24 and 48 weeks
Depression (Beck Depression Inventory-II (BDI-II)) change | 0, 24 and 48 weeks
Non-motor symptoms (Non-Motor Symptoms Questionnaire (NMSQ)) change | 0, 24 and 48 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Martin Langeskov-Christensen, Ph.d., Principal Investigator — University of Aarhus
Locations (1):
- Sport Science, Department of Public Health, Aarhus University, Aarhus, Aarhus C, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ernst M, Folkerts AK, Gollan R, Lieker E, Caro-Valenzuela J, Adams A, Cryns N, Monsef I, Dresen A, Roheger M, Eggers C, Skoetz N, Kalbe E. Physical exercise for people with Parkinson's disease: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2024 Apr 8;4(4):CD013856. doi: 10.1002/14651858.CD013856.pub3. PMID 38588457
- [Derived] Ernst M, Folkerts AK, Gollan R, Lieker E, Caro-Valenzuela J, Adams A, Cryns N, Monsef I, Dresen A, Roheger M, Eggers C, Skoetz N, Kalbe E. Physical exercise for people with Parkinson's disease: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2023 Jan 5;1(1):CD013856. doi: 10.1002/14651858.CD013856.pub2. PMID 36602886